CLINICAL TRIAL: NCT06838780
Title: Peripheral Blood Single Cell-type Expression Profile of Interferon-stimulated and Other Biomarker Genes for Triage of Febrile Patients
Brief Title: Host Response to Infection by Direct Analysis of Leukocyte Single Cell-type Gene Expression/transcript Abundance, Direct LS-TA
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Nelson Tang, Principle investigator, Chinese University of Hong Kong
Other Study IDs: Direct LS-TA retrospective
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gene Expression; Gene Expression Profiling; Infection; Viral Diseases; Bacterial Infections; Active Tuberculosis
Keywords: host response; transcriptome; Single cell-type gene expression; triage; fever; febrile patients
MeSH Terms: conditions — Infections; Virus Diseases; Bacterial Infections; Latent Tuberculosis; Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood are collected into EDTA or citrate tubes. An aliquot of whole blood (WB) will be processed for RNA fixation by addition of Trizol solution and stored in -70C before total RNA extraction. Another aliquot of WB are separated into granulocytes and PBMC by the Ficoll gradient method. Granulocytes and a portion of PBMC will be fixed by trizol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Vaccination Controls: Up to 200 adult samples collected as the baseline of this study will be used to establish the reference ranges of the ratio-based biomarkers by quantitative PCR or digital PCR.
  Interventions: Other: No intervention
- Bacterial infection samples: A retrospective sample of adult patients with positive bacterial blood culture.
  Interventions: Other: No intervention
- Tuberculosis samples: A retrospective sample of adult patients who were diagnosed to have active tuberculosis disease.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention for this retrospective study

SUMMARY:
Febrile illness is a common condition, particularly among young patients and it is crucial to have an early triage of patients according to various aetiologies to enable appropriate treatment. Most diagnostic tests are targeted towards the detection of pathogens while other assays are mostly related to serum proteins. Blood cells transcriptome has been explored to differentiate bacterial and viral infections.

Here, we propose to develop a rapid test using the host responses in terms of gene expressions of single-cell populations of peripheral leukocytes (monocytes and granulocytes) to differentiate three major categories of infections that are bacterial, viral, and tuberculosis.

The assay is called Direct leukocyte single cell-type transcript abundance (TA) assay (DIRECT LS-TA) as it can directly determine the gene expression of a specified single cell-type (e.g. monocytes and granulocytes) among various leukocyte cell populations directly in a peripheral blood sample. Such results signify the nature of host response and can be used to indicate the type of infection (viral, bacterial or active tuberculosis).

DETAILED DESCRIPTION:
DIRECT LS-TA is a ratio-based biomarker (RBB) for blood gene expression analysis which can be performed in commonly available equipments (e.g. qPCR or digital PCR machines). Using the ratio of TA of prior defined numerator gene and denominator gene, this RBB can quantify gene expression of the specified constitutional single cell-type (e.g. monocytes and granulocytes) inside a cell-mixture sample of Whole blood.

DIRECT LS-TA was a method pioneered by the PI [Tang 2017, https://patents.google.com/patent/US9589099B2/]. And it has been developed for quantification of early B cell response after vaccination [DOI: 10.3390/genes12070971].

Recently, the method is used to develop host response biomarkers after infection to differentiate the type of pathogens (such as viral, bacterial or active tuberculosis). Numerator and denominator genes have been identified by using public gene expression datasets for monocytes and granulocytes. Diagnostic performance was good using these public data.

Therefore, these RBBs will be applied in these retrospective samples to evaluate and compare their diagnostic (triage) performance of febrile patients into different pathogen etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Bacterial infection sample: positive isolation of organism in blood culture (Bacterial infection sample group)
* Clinical diagnosed active TB (Tuberculosis infection group)

Exclusion Criteria:

* End stage renal failure
* Pregnancy
* Infections for which long term antibiotic treatment is strongly recommended (including infective endocarditis, osteoarticular infections, cerebral or hepatic or lung abscesses, tuberculosis or nontuberculous mycobacterial infections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Infections were patients admitted to ward for treatment of infection.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Viral host response Direct LS-TA in monocytes (Type I interferon response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: Monocyte. RBB numerator gene: IFI27 or IFI44L. RBB denominator gene: PSAP, CTSS or CPVL.
  The various RBB (e.g. IFI27/PSAP and IFI44L/PSAP ratios) will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Viral host response Direct LS-TA in granulocytes (Type I interferon response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: Granulocyte. RBB numerator gene: RSAD2 or IFIT1. RBB denominator gene: SAT1 or SRGN.
  The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Bacterial infection host response Direct LS-TA in monocytes (pro-inflammatory response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: Monocyte. RBB numerator gene: VNN1, or NLRC4. RBB denominator gene: PSAP, CTSS or CPVL.
  The various RBBs will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Bacterial infection host response Direct LS-TA in granulocytes (pro-inflammatory response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: Granulocyte. RBB numerator gene: ALPL, ARG1, or ANXA3. RBB denominator gene: SAT1 or SRGN. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Active TB host response Direct LS-TA in monocytes (Type II interferon response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: Monocyte. RBB numerator gene: WARS1, ATF3 or CALHM6. RBB denominator gene: PSAP, CTSS or CPVL. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.
Active TB host response Direct LS-TA in granulocytes (Type II interferon response) | 1 day (first collected sample after admission)
  Direct LS-TA is a kind of RBB that can be readily quantified by qPCR or dPCR of a pair of genes, the RBB numerator gene and the RBB denominator gene. The biomarker is the ratio of the 2 genes.
  Single cell-type: granulocyte. RBB numerator gene: ANKRD22, BATF2, CD274, FCGR1A or ETV7. RBB denominator gene: SAT1 or SRGN. The various RBB will be compared in terms of their sensitivity/specificity of diagnostic performance in the vaccination control samples and samples from infection groups. AUC of ROC analysis will be performed where appropriate.

SECONDARY OUTCOMES:
Reference intervals and median of these DIRECT LS-TA RBB in the control group | 1 day (first collected sample after admission)
  The median value and the central 95% range of each RBB will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Chemical Pathology, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Descriptive statistics of each RBB (DIRECT LS-TA) will be provided on a reasonable request.

REFERENCES:
- [Background] Tang NLS, Kwan TK, Huang D, Ma SL, Leung KS. Direct single cell-type gene expression analysis in peripheral blood: novel ratio-based gene expression biomarkers using 2 novel monocyte reference genes (PSAP and CTSS) for detection of bacterial infection. Hum Mol Genet. 2025 Aug 21;34(17):1458-1470. doi: 10.1093/hmg/ddaf103. PMID 40581066
- [Background] Huang D, Liu AYN, Leung KS, Tang NLS. Direct Measurement of B Lymphocyte Gene Expression Biomarkers in Peripheral Blood Transcriptomics Enables Early Prediction of Vaccine Seroconversion. Genes (Basel). 2021 Jun 25;12(7):971. doi: 10.3390/genes12070971. PMID 34202032
- [Background] Huang B, Huang J, Chiang NH, Chen Z, Lui G, Ling L, Kwan MYW, Wong JSC, Mak PQ, Ling JWH, Lam ICS, Ng RWY, Wang X, Gao R, Hui DS, Ma SL, Chan PKS, Tang NLS. Interferon response and profiling of interferon response genes in peripheral blood of vaccine-naive COVID-19 patients. Front Immunol. 2024 Jan 10;14:1315602. doi: 10.3389/fimmu.2023.1315602. eCollection 2023. PMID 38268924
- See also: Patent about the model to obtain single cell-type gene expression in peripheral blood — https://patents.google.com/patent/US9589099B2/
- See also: Patent about the model to obtain single cell-type gene expression in peripheral blood — https://patents.google.com/patent/GB2629711A/en